CLINICAL TRIAL: NCT03901014
Title: Investigating the Production of Lipoproteins and Acetyl-CoA During a Ketogenic Diet
Acronym: PLAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Touro University, California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M-0419
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Cholesterol Metabolism; Ketone Metabolism
Keywords: ketogenic diet; LDL cholesterol; carbohydrate

STUDY DESIGN:
Masking Description: The nature of the diet does not allow for masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline diet (Active Comparator): 1 week baseline diet
  Interventions: Other: Standard American diet
- Very low carbohydrate diet (Experimental): 2 week very low carbohydrate ketogenic diet
  Interventions: Other: Very low carbohydrate diet

INTERVENTIONS:
Other: Standard American diet — Standard American diet with 50% energy from carbohydrate, 30% from fat, and 20% from protein.
  Arms: Baseline diet
Other: Very low carbohydrate diet — Ketogenic diet with <50g carbohydrate, 60-75% energy from fat, and 20% from protein
  Arms: Very low carbohydrate diet

SUMMARY:
The purpose of this study is to understand how the reduction in dietary carbohydrates in a very-low carbohydrate ketogenic diet impacts the synthesis of cholesterol, fatty acid, and ketones, and the turnover rate of VLDL and chylomicron particles.

DETAILED DESCRIPTION:
Participants will consume a standard American diet for one week followed by a very-low carbohydrate ketogenic diet (VLCKD, <50 grams carbohydrate/day) for two weeks. Participants will undergo an oral stable isotope tracer study during each diet to measure de novo synthesis of fatty acid, cholesterol, ketone bodies, and for measurement of apolipoprotein B and triglyceride kinetics.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-50 years old

Exclusion Criteria:

* Use of nicotine products
* Has dietary restrictions
* Lactose intolerance
* History of GI disorders, diabetes, liver, kidney, or thyroid disorders
* Taking hypolipidemic, anti-diabetic, anti-hypertensive, or anti-depression medication
* Screening plasma triglyceride < 50mg/dl or >500mg/dl
* Screening glucose > 125mg/dl
* Screening total and LDL-Cholesterol over 95th %tile for age and sex
* BP > 160/95 mmHg
* Weight loss/gain > 5% in the previous 3 months (self-reported)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Change in total cholesterol | Day 3-7 to Day 17-21
  Change in serum total cholesterol between Day 3-7 (average value) to Day 17-21 (average value)
Change in low density lipoprotein (LDL) cholesterol | Day 3-7 to Day 17-21
  Change in serum LDL cholesterol between Day 3-7 (average value) to Day 17-21 (average value)
Change in high density lipoprotein (HDL) cholesterol | Day 3-7 to Day 17-21
  Change in serum HDL cholesterol between Day 3-7 (average value) to Day 17-21 (average value)
Change in apolipoprotein B (apoB) kinetics | Day 3-7 to Day 17-21
  Change in apoB turnover rates in LDL and very low density lipoprotein plasma fractions as measured using 2H2 leucine incorporation into apoB and mathematical modeling

SECONDARY OUTCOMES:
Change in fractional hepatic de novo lipogenesis | Day 3 to Day 17
  Measured by the detection of incorporated 1-13C sodium acetate into palmitate in triglyceride rich lipoproteins (TRL)
Change in fractional cholesterol synthesis | Day 3 to Day 17
  Measured by the detection of incorporated 1-13C sodium acetate into cholesterol in plasma
Change in ketone body synthesis | Day 3 to Day 17
  Measured by the detection of incorporated 1-13C sodium acetate into ketone bodies in plasma
Change in TRL-triglyceride kinetics | Day 3 to Day 17
  Change in TRL- triglyceride assembly rates as measured using 2-13C glycerol and mathematical modeling
Change in triglyceride lipolysis | Day 3 to Day 17
  Measured by the dilution of administered 2-13C glycerol in plasma
Change in serum glucose concentration | Day 3 to Day 17
  Change in fasting and postprandial serum glucose levels
Change in serum free fatty acid concentration | Day 3 to Day 17
  Change in fasting and postprandial serum free fatty acid levels
Change in serum insulin concentration | Day 3 to Day 17
  Change in fasting and postprandial serum insulin levels
Change in serum ketone body concentration | Day 3 to Day 17
  Change in fasting and postprandial ketone body levels

CONTACTS AND LOCATIONS:
Overall Officials: Grace M Jones, PhD, Principal Investigator — Touro University, California
Locations (1):
- Touro University California, Vallejo, California, United States

IPD SHARING:
Plan to Share IPD: No